CLINICAL TRIAL: NCT00307112
Title: Study of the Prevalence of Rheumatic Heart Disease in Leon, Nicaragua
Brief Title: Rheumatic Heart Disease Prevalence in Leon, Nicaragua
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0093
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2011-05

CONDITIONS: Streptococcus Group A
Keywords: Group A streptococcus, Nicaragua, Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
A bacterium called Group A Steptoccoccus or "strep" is commonly found in the nose and throat of healthy adults and children and can cause a variety of illnesses. If this bacterium infects another part of the body one or more times, children may get Rheumatic heart disease (RHD). The purpose of this community based study is to see how many children between 5-15 years of age have RHD in Leon, Nicaragua. The study will also help to determine if the usual methods of detecting this disease are working. Researchers hope that this study will help to develop vaccines that may prevent "strep" infections to Nicaragua and other parts of the world. About 3,600 children will take part in the study. The children will participate for a minimum of 1 day and have a 6 month follow-up visit if they are identified as possible or probable RHD cases. Study procedures will include clinical exams and echocardiograms to determine the presence of RHD.

DETAILED DESCRIPTION:
Group A streptococcal (GrAS) infections are responsible for a wide spectrum of clinical syndromes, ranging from uncomplicated throat infections to life-threatening invasive infections. Some cases of uncomplicated and untreated pharyngitis may trigger the onset of acute rheumatic fever (ARF) accompanied by rheumatic heart disease (RHD). ARF is the most common cause of heart disease in children around the world and is associated with early morbidity and mortality. The most cost-effective method of preventing ARF and RHD would be vaccine prevention of the streptococcal infections that trigger the disease. Unfortunately, the overall burden of RHD in developing countries is unknown. This information is needed to adequately assess the potential risk- and cost-benefits of a GrAS vaccine that may eventually be introduced in countries where ARF and RHD are prevalent. The primary objective of this study is to determine the prevalence of RHD among children aged 5-15 in Leon. The secondary objective is to determine the sensitivity and specificity of clinical examination of the heart in an area of suspected high prevalence of RHD (Leon). This is an uncontrolled, observational, community-based study designed to provide detailed information about the prevalence of RHD in children in León, Nicaragua. Children and adolescents between the ages of 5 and 15 will be eligible for enrollment. Centro de Investigación en Demografía y Salud (CIDS - Center for Investigation of Demography and Health) staff will visit randomly selected dwellings with children between the target ages of 5 and 15 years, explain the nature and purpose of the study, and obtain signed informed consent from the parents or guardians of the children to collect demographic information. The study will also be discussed with all children 13 years of age or older, and their verbal agreement to participate in the study will be sought. After informed consent has been obtained and children are enrolled, CIDS staff will administer a questionnaire to capture the children's demographics. All enrolled children and their parent(s) from a given area will be offered transportation to the rheumatic heart disease clinic at HEODRA by van. CIDS staff will arrange the examinations and transportation and will inform the families appropriately. All children whose parent(s)/guardian provide informed consent will have at least one study visit at HEODRA. On the day of the scheduled clinic visit, the families will be informed again in detail about the RHD research study and written informed consent will again be obtained. All children who participate in the study will have an auscultation and a screening echocardiogram as part of the study. Those children who are identified by auscultation and/or by echocardiography to be in the "probable or possible rheumatic heart disease" groups will be asked to return for repeat echocardiography 6 months after their first examination. The primary and secondary endpoints of the study will be clinical diagnosis of RHD as confirmed by echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

All children aged 5 to 15 years of age whose parents provide consent for their study participation are eligible for this study. Children who are 13 years or older will provide verbal agreement to participate.

Exclusion Criteria:

All children 5 to 15 years old whose parents are unable or unwilling to provide informed consent and children who are 13 years or older and unable or unwilling to provide verbal agreement to study participation will not be enrolled in the study.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2193 (Actual)
Dates: Start 2006-07-13; Primary Completion 2008-11-28 (Actual); Study Completion 2008-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Escuela Oscar Danilo Rosales Arguello, León, Nicaragua